CLINICAL TRIAL: NCT05618340
Title: Pulsed Field Ablation Paroxysmal Atrial Fibrillation Using a Novel Spiral Catheter Integrated With a 3-Dimensional Mapping System: The PULSTAR Study
Brief Title: 3-Dimensional Mapping System: The PULSTAR Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shangyang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF-SYPL-003(A)
Record Dates: First submitted 2022-11-06; First posted 2022-11-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: pulse field ablation; PFA; Paroxysmal Atrial Fibrillation; PAF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, multicenter, single-group target value method study
Masking Description: Non-blind method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group target value method (Experimental): This trial is a prospective, multicenter, single-group target value method study. All subjects are treated uniformly with the pulse ablation system provided in this protocol for paroxysmal AF, and the test results for the main indicators are statistically compared with the target values, a widely accepted standard in professional medicine, and the test results are considered to be attained if the one-sided 95% confidence interval for the test results is not lower than the target values.
  Interventions: Device: Pulsed electric field ablation device;Cardiac Pulsed Electric Field Ablation Catheter

INTERVENTIONS:
Device: Pulsed electric field ablation device;Cardiac Pulsed Electric Field Ablation Catheter — Routinely placing a coronary sinus electrode catheter, puncturing the interatrial septum, placing one sheath into the left atrium, confirming that the catheter is well in place, and setting the treatment time of the pulse ablation system in advance.
  Pulmonary vein-by-pulmonary vein ablation using a circular pulse catheter, waiting for the end of the pulse ablation phase and immediate effect confirmation.

SUMMARY:
The purpose of this study is to verify the safety and efficacy of the cardiac pulse ablation system in paroxysmal atrial fibrillation to provide the basis for product registration and clinical application.

The trial will be conducted at a clinical center with appropriate clinical cases, and paroxysmal atrial fibrillation ablation procedures will be performed by an authorized investigator using the trial product. The effectiveness and safety of the cardiac pulse ablation system in the treatment of paroxysmal atrial fibrillation will be verified by collecting the treatment success rate, immediate ablation success rate, procedure time and device use evaluation within 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤75 years of age.
* Paroxysmal atrial fibrillation diagnosed by electrocardiogram or Holter ECG (including single-lead ECG recorder, lasting≥30s) within 1 year prior to enrollment.
* Clinical diagnosis of paroxysmal atrial fibrillation.
* Symptomatic patients who are ineffective or intolerant to at least one antiarrhythmic medication; or patients who are willing to undergo ablation despite not being on medication.
* Fully understand the treatment protocol and voluntarily sign the informed consent form and be willing to undergo the tests, procedures and follow-ups required by the protocol.

Exclusion Criteria:

* Patients who have undergone left atrial surgery
* Left atrial thrombosis
* Patients of childbearing age who are unable to use effective contraception during the 12-month period after enrollment
* Anterior and posterior left atrial diameter ≥ 50 mm
* Left ventricular ejection fraction (LVEF) ≤ 40%
* Previous atrial septal repair or atrial mucinous tumor
* Active implants (e.g. pacemakers, ICDs, etc.) in the body
* NYHA class III-IV cardiac function [Appendix 1]
* Clear cerebrovascular disease within the last 6 months (including cerebral hemorrhage, stroke, transient ischemic attack)
* Cardiovascular events within the last 3 months (including acute myocardial infarction, coronary intervention or heart bypass surgery, prosthetic valve replacement or repair, atrial or ventriculotomy)
* Those with acute or severe systemic infections
* Patients with severe liver or kidney disease, malignant tumors or end-stage disease that, in the opinion of the investigator, may interfere with the treatment, evaluation and compliance of this trial
* Patients with significant bleeding tendency, hypercoagulable state and severe hematologic disorders
* Patients who have participated or are participating in other clinical trials within 3 months prior to enrollment
* Patients who have other conditions that the investigator considers inappropriate for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of Treatment Success at 3-Month Post-Procedure | Refers to the postoperative phase (blank) after 3 months postoperatively
  Refers to the postoperative phase (blank) after 3 months follow-up after process, without the use of class I and class III anti-arrhythmic drugs, by ECG, Holter, or Heart rate monitoring method based on equivalent (including a single lead electrocardiogram) confirmed that there are no last 30 s or af/the room/speed events account for the number of participants into the group of the proportion of the total number.
Rate of Treatment Success at 6-Month Post-Procedure | Refers to the postoperative phase (blank) after 6 months postoperatively
  Refers to the postoperative phase (blank) after 6 months follow-up after process, without the use of class I and class III anti-arrhythmic drugs, by ECG, Holter, or Heart rate monitoring method based on equivalent (including a single lead electrocardiogram) confirmed that there are no last 30 s or af/the room/speed events account for the number of participants into the group of the proportion of the total number.
Rate of Treatment Success at 12-Month Post-Procedure | Refers to the postoperative phase (blank) after 12 months postoperatively
  Refers to the postoperative phase (blank) after 12 months follow-up after process, without the use of class I and class III anti-arrhythmic drugs, by ECG, Holter, or Heart rate monitoring method based on equivalent (including a single lead electrocardiogram) confirmed that there are no last 30 s or af/the room/speed events account for the number of participants into the group of the proportion of the total number.

SECONDARY OUTCOMES:
Immediate success rate: pulmonary vein isolation after ablation | 1 Day of surgery
  Refers to the proportion of the number of subjects electrically isolated in each AF patient after surgery to the total number of subjects enrolled. Validation was a 20-minute wait after successful electrical isolation of the pulmonary vein, followed by reconfirmation of pulmonary vein block
Evaluation of Pulse Ablation Catheter | 1 Day of surgery
  Evaluation of catheter operation performance;Catheter ablation parameters
Evaluation of Pulse Ablation equipment | 1 Day of surgery
  System software operability;System operation stability;Hardware connection validity

OTHER OUTCOMES:
The incidence of early onset (within 7 days of ablation) adverse events | Within 7 days after the surgery
  The primary safety endpoint
Incidence of adverse events and serious adverse events associated with the study device | Within 12 months after sign the informed consent form
  Secondary Security Endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, No. 83 Wenhua Road, Shenhe District, Shenyang, Liaoning Province, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No